CLINICAL TRIAL: NCT02475538
Title: Electroacupuncture for Tapering Off Long-term Benzodiazepine Use: a Randomized Controlled Trial
Brief Title: Electroacupuncture for Tapering Off Long-term Benzodiazepine Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YEUNG Wing-Fai, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AcupBen
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Benzodiazepine Dependence
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Experimental): Subjects in this group will be treated with electroacupuncture along with a gradual tapering schedule.
  Benzodiazepines will be tapered off over four weeks. The expected reduction rate of benzodiazepines should be 25% in the first two weeks and 12.5% in 3-4 days in week 3 and week 4. If the participants cannot tolerate the effects after tapering according to our suggested plan, the dose can be kept unchanged or they can reduce the dose at a slower pace.
  Subjects will receive electroacupuncture 2 times per week for 4 consecutive weeks. Electroacupuncture involves acupuncture needling at traditionally used acupoints according to Chinese medicine theory.
  Interventions: Device: Electroacupuncture
- Placebo acupuncture (Placebo Comparator): Subjects in this group will be treated with placebo acupuncture along with a gradual tapering schedule.
  Benzodiazepines will be tapered off over four weeks. The expected reduction rate of benzodiazepines should be 25% in the first two weeks and 12.5% in 3-4 days in week 3 and week 4. If the participants cannot tolerate the effects after tapering according to our suggested plan, the dose can be kept unchanged or they can reduce the dose at a slower pace.
  The subjects will be receive placebo acupuncture 2 times per week for 4 consecutive weeks. Placebo acupuncture is a treatment that simulates the procedure of acupuncture treatment but may not have the effects of acupuncture.
  Interventions: Device: Placebo acupuncture

INTERVENTIONS:
Device: Electroacupuncture — Gradual Tapering Benzodiazepines will be tapered off over four weeks. The subjects will be told by a blinded researcher to reduce their daily dose by 25% in the 1st and 2nd week. For the remaining 50%, subjects will be asked to reduce the dose by 12.5% each time for 3-4 days in the 3rd and 4th week. Subjects who are unable to taper according to the suggested plan can reduce dose at a slower pace.
  Electroacupuncture The subjects will be treated with electroacupuncture at bilateral Sishencong (EX-HN1), Anmian, Shuaigu (GB8), Touwei (ST8), Taiyang (EX-HN5), Toulinqi (GB15), Neiguan (PC6), Shenmen (HT7), Sanyinjiao (SP6), Taichong (LV3), and unilateral Yintang (EX-HN3), Shenting (GV24), and Baihui (GV20). "De qi" is achieved if possible. The intensity of electric-stimulation will be adjusted up to a level the subject can tolerate without undue discomfort. The needles will be left for 30 min.
  Arms: Electroacupuncture
Device: Placebo acupuncture — Gradual Tapering The gradual tapering procedure will be the same as in the "Electroacupuncture combined with gradual tapering" group.
  Placebo acupuncture Placebo needles designed by Streitberger will be used. The placebo needles are inserted to the site 1 inch beside the acupoints of the electroacupuncture group in order to avoid acupressure effect. The needles are held by surgical tape or hair pin to imitate the procedure of acupuncture. The needles are connected to an electric-stimulator with zero frequency and amplitude. The number, duration and frequency of treatment session will be the same as in the "Electroacupuncture combined with gradual tapering" group.
  Arms: Placebo acupuncture

SUMMARY:
This study aims to examine the efficacy of electroacupuncture for tapering benzodiazepines in long-term users. All eligible subjects will be randomized in a ratio of 1:1 to (1) Electroacupuncture combined with gradual tapering; and (2) Placebo acupuncture combined with gradual tapering.

DETAILED DESCRIPTION:
Recent randomized controlled studies support that acupuncture has beneficial effects for insomnia. Primary insomnia patients receiving electroacupuncture showed an increase in sleep diary-derived sleep efficiency from an average of 69.8% at baseline to 81.2% at 1-week post-treatment. A similar result was found in patients with residual insomnia associated with major depressive disorder.

Acupuncture is efficacious in alleviating anxiety and insomnia symptoms; hence, it may help to reduce the impacts of withdrawal symptoms during benzodiazepine tapering. However, there has been no randomized controlled trial to examine the efficacy and safety of acupuncture on benzodiazepine discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* taking benzodiazepines (World Health Organization Anatomical, Therapeutic and Chemical classification system codes N05BA, N05CD, N05CF, and M03BX07)) on more than 50% of days for at least 3 months and during their prospective 2-week record prior to baseline
* willing to withdraw their benzodiazepine use during the study,

Exclusion Criteria:

* any relapse of psychiatric disorder in the past year that required intervention,
* Hospital Anxiety and Depression Scale depression or anxiety as a tool (subscore ≥ 8) which indicates subjects with possible depression or anxiety
* have any unstable psychiatric conditions or serious physical illnesses which are judged by the investigator to render unsuitable or unsafe;
* have valvular heart defects or bleeding disorders, taking anticoagulant drugs, or are fitted with any implanted electrical device such as pacemaker, defibrillator, or brain stimulation,
* have received any acupuncture during the previous 6 months prior to baseline,
* are pregnant, breast-feeding or of childbearing potential but not using adequate contraception,
* have infection or abscess close to the site of selected acupoints and in the investigator's opinion inclusion is unsafe and
* significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (a score ≥ 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who successfully discontinued benzodiazepines | up to 12-week post-treatment

SECONDARY OUTCOMES:
The percentage of equivalent dose of benzodiazepines reduced | First week of treatment (week 1), second week of treatment (week 2), third week of treatment (week 3), fourth week of treatment (week 4), 2-week post-treatment (week 6) and 12-week post-treatment (week 16)
  Different type of benzodiazepines are tranformed into an equivalent dose of diazepam
Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ) | First week of treatment (week 1), second week of treatment (week 2), third week of treatment (week 3), fourth week of treatment (week 4), 2-week post-treatment (week 6) and 12-week post-treatment (week 16)
  20-item, self-administered withdrawal symptom questionnaire
Insomnia Severity Index (ISI) | second week of treatment (week 2), fourth week of treatment (week 4), 2-week post-treatment (week 6) and 12-week post-treatment (week 16)
  7-item 5-point Likert self-rating scale on the severity of insomnia and the distress
Hospital Anxiety and Depression Scale (HADS) | second week of treatment (week 2), fourth week of treatment (week 4), 2-week post-treatment (week 6) and 12-week post-treatment (week 16)
  14-item self-administrated questionnaire, which will be used to assess the severity of depressive and anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of Psychiatry, Kowloon Hospital, Hong Kong
  - Department of Psychiatry, Queen Mary Hospital, Hong Kong
  - Department of Psychiatry, United Christian Hospital, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Chung KF, Zhang ZJ, Zhang SP, Chan WC, Ng RM, Chan CL, Ho LM, Yu BY, Chau JC, Lau NC, Lao LX. Electroacupuncture for tapering off long-term benzodiazepine use: A randomized controlled trial. J Psychiatr Res. 2019 Feb;109:59-67. doi: 10.1016/j.jpsychires.2018.11.015. Epub 2018 Nov 22. PMID 30504097
- [Derived] Yeung WF, Chung KF, Zhang ZJ, Chan WC, Zhang SP, Ng RM, Chan CL, Ho LM, Yu YM, Lao LX. Electroacupuncture for tapering off long-term benzodiazepine use: study protocol of randomized controlled trial. BMC Complement Altern Med. 2017 Mar 31;17(1):183. doi: 10.1186/s12906-017-1692-5. PMID 28359309